CLINICAL TRIAL: NCT00260806
Title: HAART Associated Cardiotoxicity in HIV-Infected Children
Brief Title: Long-term Effects of Highly Active Anti-Retroviral Therapy on HIV-Infected Children
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Clinical Trials & Surveys Corp (C-TASC) (Industry); Baylor College of Medicine (Other); University of Illinois at Chicago (Other); Columbia University (Other); Boston Medical Center (Other); Boston Children's Hospital (Other); University of Puerto Rico (Other); State University of New York (Other)
Responsible Party: Principal Investigator, Steven E. Lipshultz, MD, Voluntary Professor, University of Miami
Other Study IDs: 1318; R01HL078522 (NIH)
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) were collected from the WITS cohort to investigate the presence of mitochondrial DNA (mtDNA) mutations.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Children perinatally infected with HIV with exposure to highly active anti-retroviral therapy (HAART).
- 2: Children with perinatally acquired HIV infection enrolled on the P2C2 Study, not exposed to HAART therapy.

SUMMARY:
This study will use the NIH-sponsored Women and Infants Transmission Study (WITS) and the Pediatric Pulmonary and Cardiovascular Complications of Vertically Transmitted HIV Infection (P2C2) HIV-infected pediatric cohorts to determine how left ventricular (LV) function (particularly fractional shortening and contractility) and structure (particularly wall thickness and mass) are affected by cumulative intensity of exposure to highly active anti-retroviral therapy (HAART).

DETAILED DESCRIPTION:
BACKGROUND:

HIV-infected children are often given HAART to reduce HIV-associated disease. The long-term effects and toxicities associated with this chronic therapy in children are unknown, but severe cardiotoxicity has been suggested in animal models.

DESIGN NARRATIVE:

The P2C2 HIV-infected pediatric cohort received non-HAART regimens in various intensities. Yet, this cohort has exhibited persistent and significant depression of LV contractility compared to uninfected children (after 5 years of follow-up). These same echocardiographic measures have proven to be independently predictive of mortality. Most of the children in the WITS HIV-infected pediatric cohort have been exposed to HAART at varying times and at varying regimen intensities. By assessing LV structure and function, with the same echocardiographic protocol in the WITS cohort as was used previously in the P2C2 cohort, the study will be able to determine the incremental effects of HAART and non-HAART regimens on LV structure and function. The study will also test the hypothesis that HAART exposure results in impaired mitochondrial function that results in cardiomyopathy. This will be assessed by comparing the parameters of LV structure and function that define cardiomyopathy to the frequency of mitochondrial DNA mutations in cells from these same patients. A nested-case-control study design of mitochondrial mutations will be used to assess the relationship between HAART, mitochondrial compromise, and LV structure and function. Treatment intensity for both HAART and non-HAART regimens will be captured through a cumulative score based on an existing 8-point ordinal scale. Intensity will be measured at three points in time: 1) in utero; 2) during the first year of life; and 3) after the first year of life. Analysis of the longitudinal echocardiographic and mitochondrial data will provide valuable information about dose intensity and the comparative impact of HAART versus less aggressive drug regimens. It will also provide information on the impact of therapy during different stages of child development. Similar longitudinal data on viral load and duration of HIV will enable the investigators to control for the effects of HIV infection on cardiovascular toxicity. The findings will help determine the need for cardiovascular follow-up, prevention, and therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children
* Mothers of children understand and are willing to provide informed consent
* Mothers of children are capable of answering in English or with the help of an interpreter

Exclusion Criteria:

* HIV-infected child who is too young (less than 2 years of age) or otherwise unable to undergo an echocardiogram without sedation
* Mothers of children have maternal diabetes or phenylketonuria
* Mothers of children have a recognized Mendelian or chromosomal defect
* Mothers of children are/were actively receiving chemotherapy for cancer during pregnancy
* Mothers of children used lithium carbonate, anticonvulsants, amphetamines, or angiotensin converting enzyme (ACE) inhibitors on a chronic basis

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study participants will be children perinatally infected with HIV who were enrolled in the Women and Infants Transmision Study (WITS).
  This cohort will be compared to the historical Pediatric Pulmonary and Cardiovacular Complications Study (P2C2 HIV) cohort of perinatally HIV-infected children not exposed to HAART.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Cardiac systolic function | Measured from 2 years of age to 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Lipshultz, MD, Principal Investigator — University of Miami
Locations (9):
- United States (8):
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Illinois - Chicago, Chicago, Illinois
  - Clinical Trials and Surveys Corp. (C-TASC), Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - State University of New York (SUNY), Brooklyn, New York
  - Columbia University, New York, New York
  - Baylor College of Medicine, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico